CLINICAL TRIAL: NCT03306771
Title: The Relationship Between Morbid Obesity and Carotid Artery Stenosis - a Comparative Prospective Study
Brief Title: The Relationship Between Morbid Obesity and Carotid Artery Stenosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Uri Kaplan , MD, MD, HaEmek Medical Center, Israel
Other Study IDs: 0126-17-EMC
Record Dates: First submitted 2017-10-01; First posted 2017-10-11 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2017-10

CONDITIONS: Carotid Artery Diseases; Morbid Obesity; Metabolic Syndrome
Keywords: Morbid Obesity; Carotid Stenosis; Metabolic Syndrome
MeSH Terms: conditions — Carotid Artery Diseases; Obesity, Morbid; Metabolic Syndrome; Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Metabolic syndrome risk factors: Candidates for bariatric surgery who have metabolic syndrome risk factors will be evaluated by Ultrasound duplex before the bariatric surgery and 6,12 and 24 months post surgery for Intimal-Media Thickness and Carotid artery velocity
  Interventions: Diagnostic Test: Ultrasound Duplex
- No metabolic Syndrome risk factors: Candidates for bariatric surgery who lack metabolic syndrome risk factors will be evaluated by Ultrasound duplex before the bariatric surgery and 6,12 and 24 months post surgery for Intimal-Media Thickness and Carotid artery velocity
  Interventions: Diagnostic Test: Ultrasound Duplex

INTERVENTIONS:
Diagnostic Test: Ultrasound Duplex — The two groups will have Ultrasound Duplex before bariatric surgery, and 6,12 and 24 months post surgery

SUMMARY:
The correlation between metabolic syndrome and carotid artery stenosis is well established. The purpose of this study is to evaluate the relationship between morbid obesity and carotid artery stenosis.

DETAILED DESCRIPTION:
The investigators hypothesis is that there is a direct relationship between morbid obesity and carotid artery stenosis. The investigators hypothesize that metabolic/Bariatric surgery improves the stenosis in the carotid artery.

This is a prospective comparative study on the candidates for metabolic/Bariatric surgery in the bariatric center, Emek Medical Center, Afula, Israel. The investigators will compare the candidate for metabolic surgery with metabolic syndrome risk factors to the ones without metabolic syndrome risk factors.

The assessment of the carotid artery will be done by Ultrasound Doppler before surgery and 6, 12 and 24 month post surgery.

ELIGIBILITY:
Inclusion Criteria:

• Candidates for first bariatric surgery

Exclusion Criteria:

* Smokers or past smokers
* Patients who are post carotid artery intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates for first bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between morbid obesity and carotid artery stenosis | 24 months post surgery
  Evaluate the correlation between the two in order to identify high risk patient for carotid stenosis without metabolic syndrome risk factors

SECONDARY OUTCOMES:
Changes in Intimal -media thickness | Before bariatric surgery, and 6,12,24 months after the surgery
  To compare the baseline Intimal-media thickness before surgery to the one post-surgery by the use of Ultrasound
Changes in the carotid artery velocity | Before bariatric surgery, and 6,12,24 months after the surgery
  To compare the baseline carotid artery velocity before surgery to the one post-surgery by the use of Ultrasound Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Uri Kaplan, MD, Principal Investigator — haemek medical center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ribeiro Filho FF, Mariosa LS, Ferreira SR, Zanella MT. [Visceral fat and metabolic syndrome: more than a simple association]. Arq Bras Endocrinol Metabol. 2006 Apr;50(2):230-8. doi: 10.1590/s0004-27302006000200009. Epub 2006 May 23. Portuguese. PMID 16767289
- [Background] Sims EA. Are there persons who are obese, but metabolically healthy? Metabolism. 2001 Dec;50(12):1499-504. doi: 10.1053/meta.2001.27213. PMID 11735101
- [Background] Sharma AM. Obesity and cardiovascular risk. Growth Horm IGF Res. 2003 Aug;13 Suppl A:S10-7. doi: 10.1016/s1096-6374(03)00047-9. PMID 12914719
- [Background] Pignoli P, Tremoli E, Poli A, Oreste P, Paoletti R. Intimal plus medial thickness of the arterial wall: a direct measurement with ultrasound imaging. Circulation. 1986 Dec;74(6):1399-406. doi: 10.1161/01.cir.74.6.1399. PMID 3536154
- [Background] Marchesi F, Giacosa R, Reggiani V, De Sario G, Tartamella F, Melani E, Mita MT, Cinieri FG, Cecchini S, Ricco' M, Salcuni P, Roncoroni L. Morphological Changes in the Carotid Artery Intima after Gastric Bypass for Morbid Obesity. Obes Surg. 2017 Feb;27(2):357-363. doi: 10.1007/s11695-016-2279-9. PMID 27389676
- [Background] Sarmento PL, Plavnik FL, Zanella MT, Pinto PE, Miranda RB, Ajzen SA. Association of carotid intima-media thickness and cardiovascular risk factors in women pre- and post-bariatric surgery. Obes Surg. 2009 Mar;19(3):339-44. doi: 10.1007/s11695-008-9783-5. Epub 2008 Dec 13. PMID 19083071